CLINICAL TRIAL: NCT05429437
Title: Assesment of Two Different Modalities of Maxillary Canine Retraction Assisted With Injectable Platelet Rich Fibrin: A Prospective Clinical Study
Brief Title: Assesment of Two Different Modalities of Maxillary Canine Retraction Assisted With Injectable Platelet Rich Fibrin
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, mohamed radwan mohamed radwan el shamy, Principal investigator, Al-Azhar University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 785/274
Record Dates: First submitted 2022-06-19; First posted 2022-06-23 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Effect of Platelet Rich Fibrin Tooth Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): will include 9 patients
  Interventions: Biological: Injectable platelet rich fibrin .
- Group II (Active Comparator): will include 9 patients.
  Interventions: Biological: Injectable platelet rich fibrin .

INTERVENTIONS:
Biological: Injectable platelet rich fibrin . — i-PRF with maxillary canine retraction that will be performed two times on intervention sides according to a standardized protocol.
  Arms: Group I
Biological: Injectable platelet rich fibrin . — i-PRF that will be performed four times on intervention sides according to a standardized protocol.
  Arms: Group II

SUMMARY:
The present prospective clinical study will be undertaken for assessment of two different modalities of maxillary canine retraction assisted with injectable platelet rich fibrin.

ELIGIBILITY:
Inclusion Criteria:

* An age range from 15-22 years.
* Severe crowding or protrusion requiring 1st premolars extractions followed by symmetrical canine retraction.
* All permanent teeth present, 3rd molars are excluded.
* Good oral and general health.
* No systemic disease/medication that could interfere with OTM. No previous orthodontic treatment.

Exclusion Criteria:

* Patient diagnosed to have an indication for non-extraction approach.
* Poor oral hygiene or periodontally compromised patient.
* Patient with craniofacial anomalies or previous history of trauma, bruxism or parafunctions.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
assessment of acceleration of canine retraction | post interventional at 4 months
  rate of canine retraction

CONTACTS AND LOCATIONS:
Overall Officials: mohamed radwan, student, Principal Investigator — Al-Azhar University
Locations (1):
- AlAzhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeitounlouian TS, Zeno KG, Brad BA, Haddad RA. Effect of injectable platelet-rich fibrin (i-PRF) in accelerating orthodontic tooth movement : A randomized split-mouth-controlled trial. J Orofac Orthop. 2021 Jul;82(4):268-277. doi: 10.1007/s00056-020-00275-x. Epub 2021 Jan 22. PMID 33481053
- [Background] Erdur EA, Karakasli K, Oncu E, Ozturk B, Hakki S. Effect of injectable platelet-rich fibrin (i-PRF) on the rate of tooth movement. Angle Orthod. 2021 May 1;91(3):285-292. doi: 10.2319/060320-508.1. PMID 33459765